CLINICAL TRIAL: NCT02165904
Title: Subarachnoid Administrations of Adults Autologous Mesenchymal Stromal Cells in Patients Suffering Incomplete Spinal Cord Injury (SCI)
Brief Title: Subarachnoid Administrations of Adults Autologous Mesenchymal Stromal Cells in SCI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Jesús Vaquero Crespo, M.D., Principal Investigator, Puerta de Hierro University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CME-LEM2; 2011-005684-24 (Registry Identifier: 2011-005684-24)
Record Dates: First submitted 2014-05-06; First posted 2014-06-18 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-05

CONDITIONS: Spinal Cord Injury
Keywords: Analyze clinical efficacy of subarachnoid administration of; autologous BMSC expanded "in vitro"
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous Mesenchymal Bone Marrow Cell (Experimental): All patients will be treated with the same treatment: Adult Autologous Mesenchymal Bone Marrow Cell
  Interventions: Biological: Adult Autologous Mesenchymal Bone Marrow Cell

INTERVENTIONS:
Biological: Adult Autologous Mesenchymal Bone Marrow Cell — Diagnosed patients with incomplete spinal cord injury and chronically established SCI will be treated with Adult Autologous Mesenchymal Bone Marrow Cells.

SUMMARY:
The study goes on 24 months, with recruiting, treatment and follow period for all patients. The first day for each patient will be the first cellular administration. 3 doses will be administrated every 3 months from first dose.

When the clinical trial finishes, it will be done a completed check of all obtained parameters.

DETAILED DESCRIPTION:
It is a clinical trial phase I, single center, non-randomized, uncontrolled, open prospective follow-up of a cohort of patients with chronic spinal cord injury (SCI) .10 patients will be included with this injury.

Primary objective: Analyze the possible clinical efficacy of administration of main adult mesenchymal autologous cells expanded "in vitro" in patients with incomplete and chronically established SCI.

Secondary objectives: Confirm the safety of treatment, and study possible changes in the cerebrospinal fluid (CSF) levels (Brain-derived neurotrophic factor (BDNF), glial cell line-derived neurotrophic factor (GDNF), nerve growth factor (NGF), ciliary neurotrophic factor (CNTF), Nerve Growth Factor 3 and 4(NT3 and NT4) after subarachnoid administration of BMMC.

ELIGIBILITY:
Inclusion Criteria:

1. Incomplete SCI
2. Neurological deficit clinically stable at least 12 months prior to treatment, and with a minimum of one-year evolution after SCI.
3. Neurophysiological confirmation of incomplete SCI.
4. The MRI study that morphologically evaluate the SCI.
5. Age between 18 and 70 years
6. Thread Men and women will compromise to use anticonceptive issues from first cell´s extraction to 6 months after last cell´s administration.
7. Ability to attend clinical follow-up and perform physical therapy through the treatment period.
8. Written and signed informed consent, according to the local regulation.
9. Hematologic and creatinin parameters, SGOT and SGPT, within the normal range, according to laboratory standards considering that small variations could be accepted based on clinical study team criteria.

Exclusion Criteria:

1. A classification in ASIA and FRANKEL clinical scales to evaluate the SCI.
2. Neurophysiological records that confirm the complete SCI.
3. Age below 18 years or above 70.
4. Pregnancy or lactation.
5. Malignancy disease diagnosed or treated within the last 5 years.
6. Patients with systemic disease that represents and additional risk to treatment.
7. Patients with uncertain commitment to follow the physical therapy and clinical visits as well as patient with a negative input in the previous phycological assessment.
8. Inability to assess the SCI features through MRI either noise due to spinal stabilization systems or any other cause.
9. Patients currently under hematopoietic growth factors treatment or who required or maintained anticoagulation.
10. Neurodegenerative disease additional.
11. History of substance abuse, psychiatric disease or allergy to the protein products used in the process of cell expansion.
12. Positive serology for HIV and syphilis.
13. Active Hepatitis B or Hepatitis C.
14. With other reason that would consider the patient ineligible for cell therapy according to the investigators judgment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesús JV Vaquero Crespo, M.D., Principal Investigator — Hospital Universitario Puerta de Hierro-Majadahonda
Locations (1):
- Hospital Puerta de Hierro, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual data of participants will be shared with Authorities at the end of the Clinical development plan by the CTD (Common Technical Document). Results will be published in a scientific publication

REFERENCES:
- [Background] Vaquero J, Zurita M. Functional recovery after severe CNS trauma: current perspectives for cell therapy with bone marrow stromal cells. Prog Neurobiol. 2011 Mar;93(3):341-9. doi: 10.1016/j.pneurobio.2010.12.002. Epub 2010 Dec 14. PMID 21163325
- [Background] Otero L, Zurita M, Bonilla C, Aguayo C, Vela A, Rico MA, Vaquero J. Late transplantation of allogeneic bone marrow stromal cells improves neurologic deficits subsequent to intracerebral hemorrhage. Cytotherapy. 2011 May;13(5):562-71. doi: 10.3109/14653249.2010.544720. Epub 2011 Jan 5. PMID 21208021

RESULTS

PARTICIPANT FLOW:
Groups:
- Autologous Mesenchymal Bone Marrow Cell: Diagnosed patients with incomplete spinal cord injury and chronically established SCI will be treated with Adult Autologous Mesenchymal Bone Marrow Cells expanded in vitro. Administrated by subarachnoid injection by lumbar puncture of 30x10^6 cells, and repeated at months 4, 7 and 10, reaching a total administration of 120x10^6 cells for each patient
Period: Overall Study
Arm/Group | Autologous Mesenchymal Bone Marrow Cell
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Autologous Mesenchymal Bone Marrow Cell
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (9.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Region of Enrollment [Number; unit: participants]
  Spain | 10

OUTCOME MEASURES:

1. Primary Outcome: Efficacy-Sensivity Improvement Using the ASIA Score
Description: Sensitivity improvement was measured using the ASIA (American Spinal Injury Association) scale to measure the Surface sensitivity (LTS), pain sensitivity (PPS), and the degree of motor function in key muscles (MS). The sum of MS, LTS, and PPS configure total ASIA score. A minimum possible score is 0 points. A maximum possible score is 224 points for a patient with normal sensation. ASIA score was obtained before surgery, and 3, 6, 9 and 12 months after surgery. Mean and standard deviation for the 10 patients were obtained at all the time points and statistically analyzed.
Time Frame: measure before treatment (baseline visit), 3, 6, 9 and 12 months after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Autologous Mesenchymal Bone Marrow Cell
Number analyzed (Participants) | 10
units on a scale
  before surgery | 188.2 (60)
  3 months | 202.2 (63.7)
  6 months | 218.4 (57.5)
  9 months | 228.9 (51.84)
  12 months | 235.5 (49.35)

2. Primary Outcome: Efficacy- Changes in Functional Independence Measure Scale
Description: - Changes in Functional Independence Measure scale (NIF scale), score at the beginning, through and the end of the treatment.
  Ranges score: 18 to 126. Being 18 total patient dependency and 126 total patient independence.
Time Frame: measure before treatment (baseline visit), 3, 6,9 and 12 months after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Autologous Mesenchymal Bone Marrow Cell
Number analyzed (Participants) | 10
score on a scale
  before surgery | 95.7 (33.9)
  3 months | 95.7 (33.9)
  6 months | 95.7 (33.9)
  9 months | 96.10 (33.42)
  12 months | 98.6 (32.05)

3. Primary Outcome: Efficacy-Change in Barthel Score
Description: - Changes in Barthel score at the beginning, through and the end of the treatment.
  Ranges score: 0 to 100. Being 0 total patient dependency and 100 total patient independence.
Time Frame: measure before treatment (baseline visit), 3, 6,9 and 12 months after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Autologous Mesenchymal Bone Marrow Cell
Number analyzed (Participants) | 10
score on a scale
  before surgery | 58 (36.07)
  3 months | 58 (36.07)
  6 months | 58 (36.07)
  9 months | 58 (36.07)
  12 months | 65 (35.59)

4. Primary Outcome: Efficacy-IANC-SCIFRS Scale
Description: -Changes in IANC-SCIFRS scale
  Ranges score: 0 to 48. Being 0 severe degree of disability and 48 normal value.
Time Frame: Changes in IANC-SCIFRS scale before surgery (baseline visit) and 3, 6, 9, 12 months after surgery (follow-up period)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Autologous Mesenchymal Bone Marrow Cell
Number analyzed (Participants) | 10
score on a scale
  before surgery | 29.10 (9.96)
  3 months | 31.5 (8.89)
  6 months | 33.90 (9.73)
  9 months | 35.9 (9.01)
  12 months | 36.9 (8.21)

5. Primary Outcome: Efficacy-Changes in PENN Score.
Description: - Changes in PENN score at the beginning, through and the end of the treatment
  Ranges score: 0 to 4. Being 0 absence of spasms and 4 frequency greater than 10 spasms per hour.
Time Frame: measure before treatment (baseline visit), 3, 6,9 and 12 months after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Autologous Mesenchymal Bone Marrow Cell
Number analyzed (Participants) | 10
score on a scale
  before surgery | 1.20 (1.14)
  3 months | 1.10 (1.10)
  6 months | 0.90 (0.88)
  9 months | 0.90 (0.88)
  12 months | 0.90 (0.88)

6. Primary Outcome: Changes in ASHWORTH Score
Description: - Changes in ASHWORTH score at the beginning, through and the end of the treatment
  Ranges score: 0 to 4. Being 0 when there isn´t increase in muscle tone when stretching, and 4 when there is rigid affected follow-up in flexion or extension
Time Frame: measure before treatment (baseline visit), 3, 6,9 and 12 months after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Autologous Mesenchymal Bone Marrow Cell
Number analyzed (Participants) | 10
score on a scale
  before surgery | 1.4 (0.81)
  3 months | 1.4 (0.81)
  6 months | 1.4 (0.81)
  9 months | 1.4 (0.81)
  12 months | 1.10 (0.99)

7. Primary Outcome: Efficacy-Changes in EVA Score
Description: • Changes in EVA score at the beginning, through and the end of the treatment
  Ranges score: 0 to 10. Being 0 absence of pain and 10 the worst pain.
Time Frame: measure before treatment (baseline visit), 3, 6,9 and 12 months after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Autologous Mesenchymal Bone Marrow Cell
Number analyzed (Participants) | 10
score on a scale
  before surgery | 1.70 (3.13)
  3 months | 0.70 (1.16)
  6 months | 0.60 (0.97)
  9 months | 0.40 (0.84)
  12 months | 0.40 (0.84)

8. Primary Outcome: Efficacy- Changes in Geffner Score
Description: changes in Geffner score before surgery (baseline visit) and 3, 6, 9, 12 months after surgery (follow-up period)
  Ranges score: 0 to 6. Being 0 absence of bladder control and 6 total control of bladder
Time Frame: Changes in Geffner scale before surgery (baseline visit) and 3, 6, 9, 12 months after surgery (follow-up period)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Autologous Mesenchymal Bone Marrow Cell
Number analyzed (Participants) | 10
score on a scale
  before surgery | 3.30 (1.34)
  3 months | 3.60 (1.26)
  6 months | 3.80 (1.14)
  9 months | 3.90 (1.10)
  12 months | 4.20 (1.23)

9. Primary Outcome: Efficacy- Changes in NBD Score
Description: changes in NBD score before surgery (baseline visit) and 3, 6, 9, 12 months after surgery (follow-up period)
  Ranges score: 0 to 47. 0-6 is very minor dysfunction. 7-9 is minor dysfunction. 10-13 is moderate dysfunction; and 14 or more is severe dysfunction.
Time Frame: measure before treatment (baseline visit), 3, 6,9 and 12 months after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Autologous Mesenchymal Bone Marrow Cell
Number analyzed (Participants) | 10
score on a scale
  before surgery | 10.60 (6.64)
  3 months | 6.10 (4.15)
  6 months | 5.70 (4.35)
  9 months | 4.40 (3.86)
  12 months | 4.20 (3.88)

10. Primary Outcome: Efficacy-Changes in the Neurophysiological Parameters (SSEPs, Somatosensory Evoked Potentials)
Description: Changes in the neurophysiological parameters (SSEPs, somatosensory evoked potentials) measured as the number of patients that improved along the study.
Time Frame: Efficacy-measure before treatment (baseline visit), 6, and 12 months after surgery
Measure: Number; unit: number of patients improved in SSEPs
Arm/Group | Autologous Mesenchymal Bone Marrow Cell
Number analyzed (Participants) | 10
number of patients improved in SSEPs
  6 months | 7
  12 months | 8

11. Primary Outcome: Efficacy-Urodynammic in Terms of Detrusor Pressure
Description: Urodynamic studies in terms of detrusor pressure (decrease on detrusor pressure is considered a clinical improvement)
Time Frame: Urodynamic studies before surgery, and at 6 and 12 months after surgery (follow-up
Measure: Mean (Standard Deviation); unit: cm/H2O
Arm/Group | Autologous Mesenchymal Bone Marrow Cell
Number analyzed (Participants) | 10
cm/H2O
  before surgery | 68.6 (20.08)
  6 months | 53.8 (20.8)
  12 months | 51.5 (37.22)

12. Primary Outcome: Efficacy-Urodynamic Studies Bladder Compliance
Description: Urodynamic studies in terms of Bladder compliance. Bladder compliance is the result of a mathematical calculation of volume responsible for 1 cm H2O pressure rise measured during a cystometric filling
  . It gives an indication on how the different mechanisms in the bladder wall react on stretching.
  It is obvious that compliance figures can vary widely in groups which makes it difficult to define limits of normality.
Time Frame: measure before treatment (baseline visit), 6 and 12 months after surgery
Measure: Mean (Standard Deviation); unit: mL/cm H2O
Arm/Group | Autologous Mesenchymal Bone Marrow Cell
Number analyzed (Participants) | 10
mL/cm H2O
  before surgery | 3.88 (3.24)
  6 months | 6.14 (3.36)
  12 months | 8.28 (6.41)

13. Primary Outcome: Efficacy-Urodynamic Studies Maximum Cystometric Capacity
Description: Urodynamic studies in terms of Maximum cystometric capacity
Time Frame: Urodynamic studies before surgery, and at 6 and 12 months after surgery (follow-up
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Autologous Mesenchymal Bone Marrow Cell
Number analyzed (Participants) | 10
mL
  before surgery | 234.9 (156.26)
  6 months | 292.4 (110.93)
  12 months | 292.6 (183.6)

14. Primary Outcome: Efficacy-modification of Magnetic Resonance Imaging (MRI)
Description: Number of patients with changes in morphology of injury compared with basal images
Time Frame: before (baseline visit) and at 12 months
Measure: Number; unit: number of patients
Arm/Group | Autologous Mesenchymal Bone Marrow Cell
Number analyzed (Participants) | 10
number of patients
  baseline | 0
  12 months | 0

15. Secondary Outcome: Number of Adverse Events .
Description: - The safety will be valued with number of adverse events related with administration of subarachnoid autologous Bone Marrow Expanded Mesenchymal Cells in Incomplete Spinal Cord Injury (SCI).
Time Frame: Up to 12 months
Measure: Number; unit: Adverse events
Arm/Group | Autologous Mesenchymal Bone Marrow Cell
Number analyzed (Participants) | 10
Adverse events | 20

16. Secondary Outcome: Efficacy- Expression of Neurotrophins in CSF (CerebroSpinal Fluid) Samples
Description: Changes in expression of neurotrophins in CSF (CerebroSpinal Fluid) samples obtained previously to first administration of cell therapy, and previously to the last administration, at month 10, in order to study the variability in the expression of neurotrophins along time. The mean+SD (standard deviation) at each time point was obtained. The tested neurotrophins were: BDNF.
Time Frame: Basal and 10 months after the administration
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Autologous Mesenchymal Bone Marrow Cell
Number analyzed (Participants) | 10
pg/ml
  BDNF before administration | 19.14 (4.58)
  BDNF in month 10 after administration | 33.82 (49.65)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Autologous Mesenchymal Bone Marrow Cell
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Mesenchymal Bone Marrow Cell (N=10)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Acute Bronchitis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Mesenchymal Bone Marrow Cell (N=10)
Hypertension (Vascular disorders) | 1 (1) — Hypertension
Local pain (General disorders) | 1 (1) — Local pain
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Leg pain
Urinary tract infection (Infections and infestations) | 2 (2) — Urinary tract infection
Headache (Nervous system disorders) | 3 (4) — Headache
Hyperthermia (General disorders) | 1 (1) — Hyperthermia
Wound (Injury, poisoning and procedural complications) | 1 (1) — Wound
Infected pressure ulcer (Infections and infestations) | 1 (1) — Infected pressure ulcer
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Arthralgia
Syncope (Nervous system disorders) | 1 (1) — Syncope
Pain in coccyx (Nervous system disorders) | 1 (1) — Pain in coccyx
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Neck pain
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Back pain
Nasopharingytis (Infections and infestations) | 1 (1) — Nasopharingytis
Bronchitis (Infections and infestations) | 1 (1) — Bronchitis
Urinary retention (Renal and urinary disorders) | 1 (1) — Urinary retention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes